CLINICAL TRIAL: NCT00045370
Title: A Phase I Study of the Safety, Tolerability, and Antitumor Activity of Escalating Doses of Intravenous CCI-779 Given in Combination With Escalating Doses of Interferon-Alpha to Patients With Advanced Renal Cancer
Brief Title: Chemotherapy and Biological Therapy in Treating Patients With Locally Advanced or Metastatic Kidney Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 02-023; CDR0000256468 (Registry Identifier: PDQ (Physician Data Query)); NCI-G02-2104; W-AR-3066K1-124-US; WYETH-C-C0125-32
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Kidney Cancer
Keywords: recurrent renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Interferon-alpha; temsirolimus

INTERVENTIONS:
Biological: recombinant interferon alfa
Drug: temsirolimus

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Biological therapies such as interferon alfa use different ways to stimulate the immune system and stop cancer cells from growing. Combining biological therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of combining chemotherapy with biological therapy in treating patients who have locally advanced or metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of CCI-779 in combination with interferon alfa in patients with locally advanced or metastatic renal cell cancer.
* Determine the safety and tolerability of this regimen in these patients.
* Determine, preliminarily, any antitumor activity of this regimen in these patients.
* Determine the pharmacokinetics of this regimen in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive interferon alfa (IFN-A) subcutaneously 3 times a week. Beginning on week 2, patients also receive CCI-779 IV over 30 minutes once weekly. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of at least 6 patients receive escalating doses of CCI-779 and then IFN-A until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, 20 additional patients are treated at that dose level.

Patients are followed at 30 days.

PROJECTED ACCRUAL: Approximately 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed locally advanced or metastatic renal cell cancer

  * Progressive disease after treatment with 0-2 courses of immunotherapy, chemotherapy, or other systemic therapy for advanced disease
* Measurable or evaluable disease
* No concurrent CNS metastases

  * Prior CNS metastases allowed if no residual disease by MRI

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 3 months

Hematopoietic

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* AST and ALT no greater than 3 times upper limit of normal (ULN) (5 times ULN if liver metastases present)

Renal

* Creatinine less than 2 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular

* No unstable angina
* No myocardial infarction within the past 6 months

Other

* Cholesterol no greater than 350 mg/dL
* Triglycerides no greater than 400 mg/dL
* HIV negative
* Not immunocompromised
* No active autoimmune disorder
* No active infection requiring antibiotic therapy
* No other serious concurrent illness
* No known hypersensitivity to components of CCI-779, interferon alfa, diphenhydramine hydrochloride, or both acetaminophen and nonsteroidal anti- inflammatory drugs
* No other major illness that would preclude study participation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* See Disease Characteristics
* At least 3 weeks since prior immunotherapy
* No prior interferon alfa
* No other concurrent immunotherapy
* No prophylactic growth factors
* Concurrent epoetin alfa allowed

Chemotherapy

* See Disease Characteristics
* At least 3 weeks since prior chemotherapy
* No prior CCI-779
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent hormonal therapy for malignancy (megestrol for appetite loss allowed)
* Concurrent inhaled or replacement steroids allowed

Radiotherapy

* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery

* At least 3 weeks since prior surgery

Other

* See Disease Characteristics
* At least 3 weeks since prior immunosuppressive agents
* At least 4 weeks since prior investigational agents
* No other concurrent investigational agents
* No concurrent immunosuppressive therapy
* No concurrent anticonvulsants known to be cytochrome P450 inducers, ketoconazole, diltiazem, rifampin, terfenadine, cisapride, astemizole, or pimozide
* No concurrent maintenance therapy for life-threatening ventricular arrhythmia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-04; Primary Completion 2003-11 (Actual); Study Completion 2003-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J. Motzer, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States